CLINICAL TRIAL: NCT00283296
Title: Development of a Collapsible Folding Manual Wheelchair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rory Cooper, Director; Pittsburgh VA Rehabilitation Research & Development Center, VA Pittsburgh Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 02331, 0408063; H133S030016
Record Dates: First submitted 2006-01-24; First posted 2006-01-27 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Wheelchair Users
Keywords: manual wheelchair; assistive technology; travel wheelchair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endeavor Wheelchair (Experimental): Participants will receive an introduction to the Endeavor wheelchair, and will complete the Activities of Daily Living Course with their own personal wheelchair and with the Endeavor chair.
  Interventions: Device: Endeavor

INTERVENTIONS:
Device: Endeavor — Collapsible, forward folding manual wheelchair

SUMMARY:
The purpose of this research study is to evaluate the Endeavor, a compact, forward-folding, ultralight manual wheelchair that incorporates small "swing-down" wheels for navigation in confined areas. This enables access to narrow environments such as those encountered in offices, restrooms, and transportation settings. When using the small access wheels, the wheelchair also fits down the aisle of airplanes and collapses to be stowed in the overhead compartment. It is anticipated that the Endeavor will maximize mobility; increase access to confined areas; and ease the demands of travel for people with disabilities.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate the Endeavor, a compact, forward-folding, ultralight manual wheelchair that incorporates small "swing-down" wheels for navigation in confined areas. This enables access to narrow environments such as those encountered in offices, restrooms, and transportation settings. When using the small access wheels, the wheelchair also fits down the aisle of airplanes and collapses to be stowed in the overhead compartment. It is anticipated that the Endeavor will maximize mobility; increase access to confined areas; and ease the demands of travel for people with disabilities.

There are two stages to this research project: an Activities of Daily Living Course and an In-Home trial. The activities of daily living course is located at the Human Engineering Research Laboratories and simulates daily barriers encountered by wheelchair users. Subjects will be asked to complete the course in their personal wheelchair and in the Endeavor three times each. Testing will be completed during a one-day visit that will not exceed 2 1/2 hours.

For the in-home trial, subjects will be asked to use the Endeavor as their primary means of mobility for two weeks, which will be compared to using their own wheelchair for two weeks. During this four-week period a datalogger will be mounted to the subject's wheelchair(s), which will give information about distance traveled, average speed, and time used. In addition to the data-logger, subjects will also be asked to keep a brief, daily, written log of the activities they performed while in the chair. At the end of the Endeavor trial-use period, subjects will be asked to complete a questionnaire. There is an 8-week follow-up period where subjects will be allowed to keep the Endeavor. We will make three calls during this period to conduct interviews on usage of the Endeavor.

ELIGIBILITY:
Inclusion Criteria:

1. Use a manual wheelchair as a primary means of mobility.
2. Male and females over the age of 18.
3. The ability to adequately fit in a wheelchair with a 16" seat width.
4. A minimum of 6 months experience using a manual wheelchair as primary means of mobility.
5. Able to transfer independently.
6. Drive own vehicle from vehicle seat.

Exclusion Criteria:

1. Active pressure sores as reported by subject.
2. History of traumatic upper extremity injury that would prevent you from folding, lifting and storing a manual wheelchair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-01; Primary Completion 2008-07 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rory A Cooper, PhD, Principal Investigator — Human Engineering Research Laboratories
Locations (1):
- Human Engineering Research Laboratories, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment and data collection occured in 2008 at the Human Engineering Research Laboratories.
Groups:
- Endeavor Wheelchair: All participants completed the Activities of Daily Living Course with their own personal wheelchair and with the Endeavor chair three times each. Testing was completed during a one-day visit that did not exceed 2 1/2 hours. For the in-home trial, subjects used the Endeavor as their primary means of mobility for two weeks and their own wheelchair for two weeks.
Period: Overall Study
Arm/Group | Endeavor Wheelchair
Started | 14
Completed | 9 (Completed in-lab and in-home trial.)
Not Completed | 5
Not completed — in-home trial not completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Endeavor Wheelchair
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reported the Endeavor to be the Same as Their Current w/c or Better With Regards to Transporting in a Vehicle
Description: Participants completed an Activities of Daily Living Course in their own personal w/c and the Endeavor. Then participants were asked to rate their level of difficulty to complete based on a 5 point likert scale: very difficult, difficult, moderate, easy, very easy. Number of participants reported the Endeavor w/c to be the same as their current w/c or better with regards to transporting in a vehicle.
Time Frame: immediately following course completion
Measure: Number; unit: participants
Groups:
- Endeavor Wheelchair: All participants received an introduction to the Endeavor wheelchair, and completed the Activities of Daily Living Course with their own personal wheelchair and with the Endeavor chair.
Arm/Group | Endeavor Wheelchair
Number analyzed (Participants) | 14
participants | 10

2. Primary Outcome: Average Distance Traveled Per/Day During the 2 Week Time Period (Personal w/c)
Description: Mean distance traveled per/day using the personal w/c was recorded with use of customized datalogger.
Time Frame: 2 week in-home trial
Population: personal w/c
Measure: Mean (Standard Deviation); unit: meters/day
Groups:
- Endeavor Wheelchair: For the in-home trial, subjects used the Endeavor as their primary means of mobility for two weeks and their own wheelchair for two weeks.
Arm/Group | Endeavor Wheelchair
Number analyzed (Participants) | 10
meters/day | 1726 (716)

3. Primary Outcome: Average Distance Traveled Per/Day During the 2 Week Time Period (Endeavor w/c)
Description: Mean distance traveled per/day using the Endeavor w/c was recorded with use of customized datalogger.
Time Frame: 2 week in-home trial
Population: Endeavor w/c
Measure: Mean (Standard Deviation); unit: meters/day
Arm/Group | Endeavor Wheelchair
Number analyzed (Participants) | 10
meters/day | 1688 (822)

ADVERSE EVENTS:
Arm/Group | Endeavor Wheelchair
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endeavor Wheelchair (N=14)
ankle/foot injury (Musculoskeletal and connective tissue disorders) | 1 — Participant bruised right foot/ankle while using the Endeavor w/c.

LIMITATIONS AND CAVEATS:
Limited number of Endeavor prototypes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No